CLINICAL TRIAL: NCT06780696
Title: Sympathetic Mapping and Ablation of Renal Nerves to Treat Uncontrolled Hypertension in Real World
Brief Title: SMART Study in Real World
Acronym: SMART-RW
Status: Not yet recruiting | Type: Observational
Sponsor: SyMap Medical (Suzhou), Ltd. (Industry)
Collaborators: Beijing Hisicom Tech Dvpt Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: SMART-RW-2024
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Uncontrolled Hypertension; Resistant Hypertension; Reduce Antihypertensive Drug Burden
Keywords: uncontrolled hypertension; hypertension; reduce antihypertensive medications; resistant hypertension
MeSH Terms: conditions — Hypertension | interventions — Radionuclide Generators

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Study: In this cohort, the long-term safety and efficacy of the approved msRDN system will be evaluated in patients with drug-resistant hypertension or patients who are intolerant to drug therapy and, in either case, need to reduce antihypertensive medications.
  Interventions: Device: SyMapCath I™ catheter and SYMPIONEER S1™ Stimulator/Generator
- Retrospective Study: In this cohort, the safety and efficacy of msRDN system will be evaluated in patients with drug-resistant hypertension or patients who are intolerant to drug therapy and, in either case, need to reduce antihypertensive medications, who have been treated by msRDN procedure.

INTERVENTIONS:
Device: SyMapCath I™ catheter and SYMPIONEER S1™ Stimulator/Generator — Radiofrequency ablation of renal arterial sympathetic nerves
  Groups: Prospective Study

SUMMARY:
This study is a multicenter, single-arm, open-label and post-market study in a real world patient population with uncontrolled hypertension to document the long-term safety and efficacy of a renal mapping/selective renal denervation (msRDN) system (SyMap Medical (Suzhou), Ltd, Suzhou, China) and conducted in accordance with the requirements by National Medical Production Administration (NMPA) of China. The msRDN system consists of a disposable renal artery radiofrequency ablation catheter (Registration No: National Medical Device Approval 20243011383), a console with both electronic stimulation and radiofrequency ablation function (Registration No: National Medical Device Approval 20243011384). The study includes prospective cohort and retrospective cohort.

Approximately1,000 patients with uncontrolled hypertension who undergo msRDN procedure will be recruited from over 30 centers in China. Subjects enrolled in the study will be followed for at least three years after msRDN procedure. This study includes patients with drug-resistant hypertension or patients who are intolerant to drug therapy and, in either case, need to reduce antihypertensive medications per the inclusion criteria defined in the protocol.

DETAILED DESCRIPTION:
A. **Prospective Study: ** In this cohort, the long-term safety and efficacy of the approved msRDN system will be evaluated in patients with drug-resistant hypertension or patients who are intolerant to drug therapy and, in either case, need to reduce antihypertensive medications.

Study Period and Timeline (for A. Prospective Cohort)**

Subjects included in this post-market, real-world study will be followed for at least three years after msRDN procedure. The regarding clinical parameters will be taken at baseline and at each follow-up as below:

* Visit 0: Baseline/Screening Period
* Visit 1: msRDN procedure (Day 0)
* Visit 2: 1 Month Post-msRDN (30 ± 7 days)
* Visit 3: 3 Months Post-msRDN (90 ± 14 days)
* Visit 4: 6 Months Post-msRDN (180 ± 30 days)
* Visit 5: 12 Months Post-msRDN (360 ± 30 days)
* Visit 6: 24 Months Post-msRDN (720 ± 30 days)
* Visit 7: 36 Months Post-msRDN (1080 ± 30 days)

B. **Retrospective Study:** In this cohort, the safety and efficacy of msRDN system will be evaluated in patients with drug-resistant hypertension or patients who are intolerant to drug therapy and, in either case, need to reduce antihypertensive medications, who have been treated by msRDN procedure.

*Study Period and Timeline (for B. Retrospective Cohort) ** Patients who have been consented and enrolled in the study will be followed for at least three years.

In this cohort, as long as a patient meets inclusion criteria of the study and at least one clinical efficacy endpoint is recorded at ≥36 months after msRDN procedure, the data from this patient will be used for statistical analysis. During 36 month study period, data will be collected at baseline and at each follow-up point per protocol as below:

* Visit 1: msRDN procedure (Day 0)
* Visit 2: 1 Month Post-msRDN (30 ± 14 days)
* Visit 3: 3 Months Post-msRDN (90 ± 28 days)
* Visit 4: 6 Months Post-msRDN (180 ± 28 days)
* Visit 5: 12 Months Post-msRDN (360 ± 28 days)
* Visit 6: 24 Months Post-msRDN (720 ± 28 days)
* Visit 7: 36 Months Post-msRDN (1080 ± 28 days) Final Follow-Up

The midpoints of two adjacent follow-ups are used as the reference to determine which follow-up point the data belong to: if data are collected before the midpoint and accounted in the early follow-up；if data are collected after the midpoint and accounted in the later follow-up.

ELIGIBILITY:
1. **Inclusion Criteria (for A. Prospective Cohort)**

   * Patients are ≥18 years old;
   * Patients with drug-resistant hypertension patients who are intolerant to drug therapy and, in either case, need to reduce medications;
   * Patients consent to receive msRDN treatment using the commercially available msRDN system by SyMap Medical (Suzhou), Ltd and to fulfill follow-up requirements.
2. **Exclusion Criteria (for A. Prospective Cohort)**

   * Subjects are withdrawn from the study due to various reasons;
   * Investigators, ethics committees or regulatory agencies may halt or terminate the study due to medical perspectives or ethical considerations.
3. **Inclusion Criteria (for B. Retrospective Cohort)**

   * Patients are ≥18 years old;
   * Patients with drug-resistant hypertension patients who are intolerant to drug therapy and, in either case, need to reduce medications;
   * Patients who have been received msRDN procedure using commercially available msRDN system by SyMap Medical (Suzhou), Ltd;
4. **Exclusion Criteria (for B. Retrospective Cohort) **

   * Subjects are withdrawn from the study due to various reasons;
   * Investigators, ethics committees or regulatory agencies may halt or terminate the study due to medical perspectives or ethical considerations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing renal denervation procedure for hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Office systolic blood pressure (OSBP) | 6 months
  The change in office systolic blood pressure between baseline and 6 months

SECONDARY OUTCOMES:
Office Blood Pressure | 1, 3, 6 (diastolic blood pressure), 12, 24 and 36 months
  Changes in office blood pressure (systolic and diastolic) between baseline and 1, 3, 6 (diastolic blood pressure), 12, 24 and 36 months, respectively;
24-hour Ambulatory Blood Pressure | 1, 3, 6, 12, 24 and 36 months
  Changes in 24-hour ambulatory blood pressure (systolic and diastolic) between baseline and 1, 3, 6, 12, 24 and 36 months, respectively;
Change in Antihypertensive Medications | 1, 3, 6, 12, 24 and 36 months
  Changes in antihypertensive medications between baseline and 1, 3, 6, 12, 24 and 36 months, respectively;
Renal Function (eGFR and UACR) | 1, 3, 6, 12, 24 and 36 months
  Changes in renal function (eGFR and UACR) between baseline and 1, 3, 6, 12, 24 and 36 months, respectively;
Blood Glucos | 1, 3, 6, 12, 24 and 36 months
  Changes in blood glucose level between baseline and 1, 3, 6, 12, 24 and 36 months, respectively

OTHER OUTCOMES:
Success rate of msRDN procedure | During the procedure
  The success rate was defined by whether the renal mapping/denervation catheter can be engaged in the correct position in the renal artery and renal nerve ablation procedure was successfully performed without related complications such as renal arterial perforation or renal artery embolization.
Success rate of clinical treatment | wiwithin 7 days after the procedure or at the time the patient is discharged from hospital
  Based on succeed performance of msRDN procedure, there are no the procedure-related SAE, such as acute infection and renal dysfunction
All-cause mortality and incidence of severe renal function impairment | 1, 3, 6, 12, 24 and 36 months
  eGFR < 15 mL/min/m² or requiring renal replacement therapy at 1, 3, 6, 12, 24 and 36 months after msRDN procedure;
Incidence of renal artery stenosis | 12, 24 and 36 months
  Incidence of renal artery stenosis (stenosis>70%) at 12, 24 and 36 months after msRDN procedure;
Incidence of adverse events | 1, 3, 6, 12, 24 and 36 months
  Incidence of adverse events and serious adverse events at 1, 3, 6, 12, 24 and 36 months after msRDN procedure.

CONTACTS AND LOCATIONS:
Overall Officials: JianPing LI, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No